CLINICAL TRIAL: NCT01828957
Title: Randomized, Double-blind, Multi-center, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Pneumostem® Versus a Control Group for Treatment of Bronchopulmonary Dysplasia in Premature Infants
Brief Title: Efficacy and Safety Evaluation of Pneumostem® Versus a Control Group for Treatment of BPD in Premature Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-CR-009
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2017-04

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Human Umbilical Cord Blood Derived Mesenchymal Stem Cells; Bronchopulmonary dysplasia; Premature infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pneumostem® (Experimental): A single intratracheal administration of Pneumostem® (1.0 x 10^7 cells/kg)
  Interventions: Biological: Pneumostem®
- normal saline (Placebo Comparator): A single intratracheal administration of normal saline
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: Pneumostem®
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: Pneumostem®
Other: Normal Saline
  Arms: normal saline

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of a single intratracheal administration of Pneumostem® for treatment of Bronchopulmonary Dysplasia (BPD) in high-risk premature infants by comparing Pneumostem-treated group with a control group.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5 - 14 days since birth
* Fetal gestational age: ≥23 weeks and <29 weeks
* Birth weight: ≥500g and ≤1250g
* Premature infant of equal to or less than 2 weeks of age who is receiving a ventilator therapy at a rate of > 12 breath/min and > 25% oxygen
* Patient whose ventilator setting has not been changed and who has shown aggravation of the illness within the 24 hours prior to the study enrollment
* Patient with a written consent form signed by a legal representative or a parent upon explanation of the clinical trial

Exclusion Criteria:

* Patient with concurrent cyanotic or acyanotic congenital heart diseases, except for patent ductus arteriosus
* Patient with a concurrent severe lung malformation (i.e. Pulmonary hypoplasia, congenital diaphragmatic hernia, congenital cystic lung disease)
* Patient with a concurrent severe lung malformation with chromosome anomalies (i.e. Edward syndrome, Patau syndrome, Down syndrome, etc) or severe congenital malformation (Hydrocephalus, Encephalocele, etc)
* Patient with a concurrent severe congenital infection (i.e. Herpes, Toxoplasmosis, Rubella, Syphilis, AIDS, etc)
* Patient withCRP > 30 mg/dL; Severe sepsis or shock
* Patient who is scheduled for or expected to undergo a surgical procedure 72 hours prior to/following the administration of the study drug
* Patient who has been administered with a surfactant within the 24 hours prior to the administration of the study drug
* Patient with severe intracranial hemorrhage ≥ grade 3 or 4
* Patient with active pulmonary hemorrhage or active air leak syndrome at the time of screening
* Patient with a history of participating in other clinical studies
* Patient who is allergic to Gentamicin
* Patient who is considered inappropriate to participate in the study by the investigator

Ages: 5 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of BPD (moderate to severe) or mortality at 36 weeks PMA | 36 weeks PMA
  Incidence of BPD (moderate to severe) or mortality rate at 36 weeks PMA

SECONDARY OUTCOMES:
Intubation duration | 36 weeks PMA
Incidence of BPD | 28-days since birth
Survival rate | 28-days since birth, 36 weeks PMA, and termination of the trial
Duration of ventilator dependence | Week 24
Duration of CPAP treatment | Week 24
Postnatal steroid use (%) for the purpose of ventilator weaning | Week 24
Cumulative duration of oxygen use | Week 24
Incidence of Retinopathy of Prematurity (ROP) of Grade III or more | Week 24
Retinopathy of Prematurity (ROP) that require treatment with avastin or laser | Week 24
Growth velocity (Z-score) | Week 24
Length of stay prior to the first discharge from the hospital | duration of the hospital stay, an expected average of approximately 3 months since birth
Incidence of adverse events | Week 24
Clinically significant laboratory findings | Week 24
Incidence of pneumothorax that require intubation | Week 24
Incidence of moderate to severe pulmonary hemorrhage | Week 24
Incidence of intraventricular hemorrhage of grade 3 or more | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Won-Soon Park, MD, PhD, Principal Investigator — Department of Pediatrics, Samsung Medical Center; Ai-Rhan Kim, Principal Investigator — Department of Neonatology, Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Ahn SY, Chang YS, Lee MH, Sung SI, Lee BS, Kim KS, Kim AR, Park WS. Stem cells for bronchopulmonary dysplasia in preterm infants: A randomized controlled phase II trial. Stem Cells Transl Med. 2021 Aug;10(8):1129-1137. doi: 10.1002/sctm.20-0330. Epub 2021 Apr 20. PMID 33876883
- See also: Related Info — http://clinicaltrials.gov/ct2/show/NCT01297205?term=medipost&rank=2